CLINICAL TRIAL: NCT02594319
Title: Understanding Mechanisms of Health Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Angela Bryan, PI, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14-0684
Record Dates: First submitted 2015-10-30; First posted 2015-11-03 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Fruit and Vegetable Consumption; Incentive Interventions
MeSH Terms: interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Daily reporting of fruit and vegetable consumption
  Interventions: Behavioral: Self monitoring
- Daily reward (Experimental): Incentives for fruit and vegetable consumption delivered daily
  Interventions: Behavioral: Monetary incentives; Behavioral: Self monitoring
- Delayed reward (Experimental): Incentives for fruit and vegetable consumption delivered in a lump sum at the end of the intervention
  Interventions: Behavioral: Monetary incentives; Behavioral: Self monitoring

INTERVENTIONS:
Behavioral: Monetary incentives
  Arms: Daily reward; Delayed reward
Behavioral: Self monitoring

SUMMARY:
This research seeks to examine psychological factors that may impact relationship between incentives and health behavior engagement, specifically fruit and vegetable consumption. Additionally, it will compare the impact of two different incentive schedules on behavior engagement, one providing immediate rewards (i.e. rewards received on a daily basis) and another providing delayed rewards (i.e. rewards received at the end of the study period), with a control condition in which no rewards are offered. Study participants will provide reports of their fruit and vegetable consumption each day for three weeks, and in the two incentive conditions, they will receive small monetary rewards for their fruit and vegetable consumption. Following the three week reporting and reward period, participants will complete two additional assessments, measuring psychological constructs and behavior engagement following the cessation of rewards.

ELIGIBILITY:
Inclusion Criteria:

* Consume fewer than 5 servings/day of fruits and vegetables
* Daily access to internet for 3 weeks following baseline session
* Have or are willing to create an account on PayPal

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Fruit and Vegetable Consumption, servings per week | 3 weeks
Perceived Behavioral Control scale score | 3 weeks
Attitudes scale score | 3 weeks
Intrinsic Motivation scale score | 3 weeks
Fruit and vegetable consumption, servings per week | 5 weeks
Perceived Behavioral Control scale score | 5 weeks
Attitudes scale score | 5 weeks
Intrinsic Motivation scale score | 5 weeks

SECONDARY OUTCOMES:
Perceived Stress Scale score | 3 weeks
Perceived Stress Scale score | 5 weeks

REFERENCES:
- [Derived] Gardiner CK, Bryan AD. Monetary Incentive Interventions Can Enhance Psychological Factors Related to Fruit and Vegetable Consumption. Ann Behav Med. 2017 Aug;51(4):599-609. doi: 10.1007/s12160-017-9882-4. PMID 28176150